CLINICAL TRIAL: NCT03416582
Title: Feasibility Study of a Nurse-Delivered Telephone Intervention To Impact Mucositis Symptom Severity and Prevent Dehydration in Lung and Head/Neck Cancer Patients Undergoing Chemoradiation: A Pilot Study
Brief Title: Feasibility Study of a Nurse Intervention to Impact Mucositis Severity and Prevent Dehydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Raphael Yechieli, Associate Professor of Clinical Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180475
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer; Mucositis Oral; Dehydration; Head and Neck Cancer
MeSH Terms: conditions — Lung Neoplasms; Stomatitis; Dehydration; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMENC Group (Experimental): The Symptom Management Education and Nurse Coaching (SMENC) intervention is a one hour in-person face-to-face education session followed by twice weekly telephone calls conducted all throughout the patient's chemoradiation treatment regimen.
  During the telephone call, the patient will report the use of the Drinks Diary.
  Interventions: Behavioral: Symptom Management Education and Nurse Coaching; Behavioral: Drinks Diary

INTERVENTIONS:
Behavioral: Symptom Management Education and Nurse Coaching — The registered nurse (RN) will teach good mouth care and management of sore mouth or throat (mucositis) symptoms to the patient for self-management at home. The RN will then call the patient twice every week to continue educating and coaching the patient about the mucositis self-management. The patient will receive the Symptom Management (SxM) Toolkit which is a written educational guide known as the "Cancer Treatment Symptom Management Education Toolkit" geared to help the patient manage their symptoms of sore mouth and throat at home in order to prevent dehydration.
Behavioral: Drinks Diary — The patient will complete the Drinks Diary daily by recording the all oral fluid ingested and also record the number of times the bathroom is used.

SUMMARY:
This is a descriptive mixed method pilot study to determine the feasibility of a tailored nurse-delivered telephone intervention designed to impact mucositis symptom severity and prevent dehydration in lung and head/neck cancer patients undergoing chemoradiation, therefore reducing overall symptom severity and improving quality of life. Secondary purposes for this study are to investigate if the nursing intervention can decrease lung and head/neck cancer patients' unscheduled medical visits between chemoradiation treatments.

ELIGIBILITY:
Inclusion Criteria:

* Non-Small Cell or Limited Stage Small Cell Lung Cancer OR Head & Neck Cancer
* Over 18 years old
* Eligible for concurrent Chemoradiation in the first line setting
* Eastern Cooperative Group 0-2 (able to complete Activity of Daily Living (ADLs) independently or with assistive device only)
* Able to read & write English or Spanish

Exclusion Criteria:

* Under 18 years old
* Underlying Anxiety or Depression (must pass screening tools)
* Medically Diagnosed with a Cognitive Impairment
* No prior Chemotherapy or Radiation treatment
* No access to a telephone
* Blind or Deaf or Illiterate
* Requires assistance with Self-Care ADLs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Number of participants that completed calls | 6 weeks
  Defined as the number of participants that completed 80% of the total 12 calls.
Duration of phone call | 6 weeks
  Amount of time of the patient daily phone call (in minutes).
Percentage of patients using Intervention materials | 6 weeks
  Percentage of the patients who reports using the interventions materials (SxM Toolkit and Drinks Diary).

SECONDARY OUTCOMES:
Attrition Rate | 6 weeks
  Attrition rate will be comprised of those study participants who drop out of the study and be computed as a percent.
Study Completion Rate | 6 weeks
  Length of time spent in the study will be expressed as a percent and it is expected that the participants will complete 75% of their planned chemoradiation treatments.
Participant Satisfaction | 6 weeks
  Qualitative analysis of a customized Semi-Structured Interview
Change in severity of mucositis | 6 weeks
  Mucositis severity will be measured daily by the Oral Mucositis Daily Questionnaire (OMDQ).
  A score of 0 equals no mucositis severity and high mucositis severity equals a score of 4 on question 2.
Change in overall symptom severity | 10 weeks
  The M.D. Anderson Symptom Inventory - Lung Cancer / Head & Neck Cancer(MDASI-LC; MDASI-HN) will be used to measure overall severity.
  The total MDASI-LC; HN score will be used in the analysis of overall symptom severity. Friedman's test is the test statistic that will be used to measure the effect of the intervention on overall symptom severity per cycle of chemoradiation treatment.
Change in quality of life | 10 weeks
  Health Related Quality of Life (HRQoL) will be measured by the Functional Assessment of Cancer Therapy - Lung and Head & Neck versions (FACT-L; FACT-H&N respectively ). The FACT-L & FACT H&N are both a five domain, 36 item self-report instrument scored on a 5 point Likert scale (zero to 4) with a score range of 0-144; the higher the score = higher HRQoL.
Unscheduled Medical Visits | 6 weeks
  Number of unplanned medical visits made by the patient to the Oncologist for intravenous fluid administration.
Influence of Nurse-Delivered Telephone Intervention on Self-Efficacy | 10 weeks
  The adapted Chronic Disease Self-Efficacy Scale (CDSES) was developed by combining the subscales of Manage Disease in General Scale and the Symptoms Scale for a combined 10 item scale to measure the concept of perceived self-efficacy. Each item is scored 0 to 8; with the higher combined sum score equating to a higher perceived self-efficacy in the participant.
Influence of Nurse-Delivered Telephone Intervention on Symptom Self-Management | 10 weeks
  The Partners in Health Scale (PIHS) was designed to measure adherence to treatment, knowledge of disease, management of side effects and management of signs and symptoms over time. The 12 item questionnaire scores each question among the domain categories on a 9 point scale from 0-8 and the higher sum score reflects a higher self-management in the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Yechieli, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Cancer Center, Miami, Florida, United States